CLINICAL TRIAL: NCT05067101
Title: A Randomized Controlled Study to Compare the Oncology Outcome and Functional Recovery of Capsule Sparing Cystectomy and Radical Cystoprostatectomy with Detaenial Sigmoid Neobladder in Men Suffering from Bladder Cancer
Brief Title: Comparison Capsule Sparing Cystectomy and Radical Cystoprostatectomy in Men with Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Chunxiao Liu, Professor;Chief Surgeon, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJH-CSC003
Record Dates: First submitted 2021-09-22; First posted 2021-10-05 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; detaenial sigmoid neobladder; prostate capsule sparing
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capsule Sparing Cystectomy (Experimental): Patients undergoing transurethral resection and enucleation of the prostate before laparoscopic cystectomy
  Interventions: Procedure: Capsule Sparing Cystectomy (CSC)
- Conventional Radical Cystoprostatectomy (Placebo Comparator): Patients undergoing conventional radical cystoprostatectomy
  Interventions: Procedure: Conventional Radical Cystoprostatectomy (CRC)

INTERVENTIONS:
Procedure: Capsule Sparing Cystectomy (CSC) — Adopt endoscopic enucleation technology to preserve the prostate capsule and part of the urinary control support structure to help restore urinary control and erectile functions
  Arms: Capsule Sparing Cystectomy
Procedure: Conventional Radical Cystoprostatectomy (CRC) — According to the consensus standard program, remove the accessory tissues including the bladder, prostate and seminal vesicles
  Arms: Conventional Radical Cystoprostatectomy

SUMMARY:
Bladder cancer is a common malignant tumor of the urinary system, radical resection plus urinary diversion is the first choice of treatment for muscle invasive bladder cancer. Urinary diversion of surgical options related to patient'survival and quality of life.

In 2000, professor Chunxiao Liu invented "detaenial sigmoid neobladder", this surgical method overset the traditional intestinal detubularization approach, which detached the serosal layer with smooth muscle from the bowel without split it. This kind of neobladder is easier to construct and have less impact on intestinal function. So far, it has been implemented for more than 700 cases in Zhujiang hospital, the age of patients range from 9 months (bladder rhabdomyosarcoma) to 88 years old.

The filed of standard radical bladder cancer resection includes the structure of the prostate and seminal vesicles. More and more studies and long-term clinical experience in our hospital have confirmed that capsule sparing cystectomy can achieve good tumor control and excellent functional recovery.

Our project is going to perform a randomized controlled trial for capsule sparing cystectomy and conventional radical cystoprostatectomy and look forward to assess the oncology outcome and functional recovery of these two procedures which provide an objective basis for the patients undergoing orthotopic urinary diversion in the future.

DETAILED DESCRIPTION:
CSC group：patients undergoing transurethral resection and enucleation of the prostate first, do not open the bladder neck to maintain the integrity of the bladder neck. The enucleated prostate capsule is preserved under laparoscopic surgery, and the urinary catheter is stretched during the operation to avoid implantation and metastasis.

CRC group：patients undergoing conventional radical cystoprostatectomy. All the patients undergoing detaenial sigmoid neobladder after cystectomy and accept at least 36 months follow up.

Followup: Patients were followed up at every 3-6 mo after surgery in the first 2 yr. The last follow-up was in the 36th month. Biochemical examination、blood and urine routine tests were done every 3 to 12 months. Urodynamic investigation, cystoscopic examination, pelvic computerized tomography, renal dynamic imaging and retro-cystogram were also performed every 3 to 12 months postoperatively.

Postoperative complications were classified as early (90 days or less) and late (greater than 90 days). Early and late complications were subdivided into those related and not related to the neobladder. Complication grade was classified according to the Clavien-Dindo system. Major complications were defined as grade III or higher.

During the follow-up period, patients were asked about daytime and night-time continence and erectile function (EF). Bladder Cancer Index and International Index of Erectile Function-5 (IIEF-5) are designed to evaluate patients' urinary control and sexual function

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 and above and healthy volunteers are not accepted;
* Bladder carcinoma in situ、T1G3 tumor、muscle invasive bladder cancer with clinical stage of cT2-T3N0M0 (If the clinical staging before neoadjuvant therapy meets the inclusion criteria, patients who have decreased to below cT2 after neoadjuvant therapy can also choose to be included according to the patient's wishes).
* Recurrent bladder cancer: recurrent NMIBC after treatment and Carcinoma in situ that does not respond to BCG vaccine treatment.
* ECOG score is 0 or 1.
* Voluntarily signed the informed consent.

Exclusion Criteria:

* Preoperative serum creatinine more than 2.26mg/dl Or 200μmol/L.
* Cancer invaded prostate or urethral (confirmed by the pathology).
* Patients with distant metastasis.
* Abnormal PSA level, or suspected patients with unconfirmed prostate cancer .
* A history of other malignant tumors within three years.
* sigmoid chronic inflammation, like ulcerative colitis or intestinal tuberculosis, and so on.
* Severe cardiopulmonary and liver dysfunction, combined with other serious diseases
* Other conditions that have been approved by a urologist for not suitable for neobladder surgery.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only male patient have prostate
Enrollment: 126 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative urinary function | At the 12th month after surgery
  Assess post-operative urinary function using the bladder cancer index (BCI) at the 12th month after surgery

SECONDARY OUTCOMES:
bladder cancer specific survival rate | 36 months
  Determine bladder cancer control with CSC compared to CRC as measured by margin status and time to disease recurrence
Sexual function | 36 months
  Assess post-operative sexual function using IIEF-5 score
Intraoperative conditions | 24 hour
  Including surgical time, bleeding volume, blood transfusion volume, etc.
Early postoperative rehabilitation indicators | 30 days after surgery
  Including intensive care time, time to restore full flow diet, hospitalization time, drainage tube removal time, visual pain score, etc
Rate of serious complications | 36 months
  Assess rate of serious complications using Clavien Dindo Complication Grading System

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiao Liu, doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Chunxiao Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Witjes JA, Bruins HM, Cathomas R, Comperat EM, Cowan NC, Gakis G, Hernandez V, Linares Espinos E, Lorch A, Neuzillet Y, Rouanne M, Thalmann GN, Veskimae E, Ribal MJ, van der Heijden AG. European Association of Urology Guidelines on Muscle-invasive and Metastatic Bladder Cancer: Summary of the 2020 Guidelines. Eur Urol. 2021 Jan;79(1):82-104. doi: 10.1016/j.eururo.2020.03.055. Epub 2020 Apr 29. PMID 32360052
- [Background] Xu K, Liu CX, Zheng SB, Li HL, Xu YW, Xu AB, Chen BS, Shen HY. Orthotopic detaenial sigmoid neobladder after radical cystectomy: technical considerations, complications and functional outcomes. J Urol. 2013 Sep;190(3):928-34. doi: 10.1016/j.juro.2013.03.072. Epub 2013 Mar 26. PMID 23538237
- [Background] Xu A, Li B, Li H, Zheng S, Du W, Xu Y, Zou Y, Luo Q, Liu C. Comparison of seromuscular tunnel and split-cuff nipple antireflux ureteroenteral anastomosis techniques in orthotopic taenia myectomy sigmoid neobladder: a prospective, randomized study. Urology. 2013 Mar;81(3):669-74. doi: 10.1016/j.urology.2012.11.018. Epub 2013 Jan 3. PMID 23290142
- [Background] Xu P, Chen C, Chen B, Bi E, Du W, Jiang N, Liu Z, Lan H, Cao M, Liu Y, Huang J, Shen H, Liu C, Liu C, Xu A. Long-term Follow-up of Detaenial Sigmoid Neobladder Reconstruction for Paediatric Patients with Bladder and Prostate Rhabdomyosarcoma: Technique and Results from a Single High-volume Centre. Eur Urol. 2022 Nov;82(5):543-550. doi: 10.1016/j.eururo.2022.08.015. Epub 2022 Aug 30. PMID 36050131
- [Background] Jacobs BL, Daignault S, Lee CT, Hafez KS, Montgomery JS, Montie JE, Humrich JE, Hollenbeck BK, Wood DP Jr, Weizer AZ. Prostate capsule sparing versus nerve sparing radical cystectomy for bladder cancer: results of a randomized, controlled trial. J Urol. 2015 Jan;193(1):64-70. doi: 10.1016/j.juro.2014.07.090. Epub 2014 Jul 24. PMID 25066875
- [Background] Hernandez V, Espinos EL, Dunn J, MacLennan S, Lam T, Yuan Y, Comperat E, Cowan NC, Gakis G, Lebret T, van der Heijden AG, Witjes JA, Ribal MJ. Oncological and functional outcomes of sexual function-preserving cystectomy compared with standard radical cystectomy in men: A systematic review. Urol Oncol. 2017 Sep;35(9):539.e17-539.e29. doi: 10.1016/j.urolonc.2017.04.013. Epub 2017 May 8. PMID 28495555
- [Background] Liu C, Zheng S, Li H, Xu K. Transurethral enucleation and resection of prostate in patients with benign prostatic hyperplasia by plasma kinetics. J Urol. 2010 Dec;184(6):2440-5. doi: 10.1016/j.juro.2010.08.037. Epub 2010 Oct 16. PMID 20952005
- [Background] Chen P, Xu P, Liu C. Long-term outcomes of bipolar transurethral enucleation and resection of the prostate on patients with benign prostatic obstruction: a 10-year follow-up. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2023 Dec;167(4):340-346. doi: 10.5507/bp.2022.034. Epub 2022 Jul 18. PMID 35938386
- [Background] Gilbert SM, Wood DP, Dunn RL, Weizer AZ, Lee CT, Montie JE, Wei JT. Measuring health-related quality of life outcomes in bladder cancer patients using the Bladder Cancer Index (BCI). Cancer. 2007 May 1;109(9):1756-62. doi: 10.1002/cncr.22556. PMID 17366596
- [Background] Gilbert SM, Dunn RL, Hollenbeck BK, Montie JE, Lee CT, Wood DP, Wei JT. Development and validation of the Bladder Cancer Index: a comprehensive, disease specific measure of health related quality of life in patients with localized bladder cancer. J Urol. 2010 May;183(5):1764-9. doi: 10.1016/j.juro.2010.01.013. Epub 2010 Mar 17. PMID 20299056
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912